CLINICAL TRIAL: NCT04581174
Title: Effect of Extraesophageal Reflux on Inferior Nasal Turbinates Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: University Hospital Bratislava (Other); Fortmedica Prague (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-turbinates_hypertrophy
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Inferior Nasal Turbinate Hypertrophy; Extraesophageal Reflux
Keywords: Inferior nasal turbinate hypertrophy; Extraesophageal reflux; Oropharyngeal pH monitoring; Restech system
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled to a total of four study arms, depending on the degree of inferior turbinates hypertrophy (according to Camacho)
Masking Description: No masking is being used in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1st degree of hypertrophy according to Camacho (Experimental): Patients with 1st degree of hypertrophy according to Camacho will undergo 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated.
  Interventions: Diagnostic Test: 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated
- 2nd degree of hypertrophy according to Camacho (Experimental): Patients with 2nd degree of hypertrophy according to Camacho will undergo 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated.
  Interventions: Diagnostic Test: 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated
- 3rd degree of hypertrophy according to Camacho (Experimental): Patients with 3rd degree of hypertrophy according to Camacho will undergo 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated.
  Interventions: Diagnostic Test: 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated
- 4th degree of hypertrophy according to Camacho (Experimental): Patients with 4th degree of hypertrophy according to Camacho will undergo 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated.
  Interventions: Diagnostic Test: 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated

INTERVENTIONS:
Diagnostic Test: 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated — Patients with the 1st degree of hypertrophy according to Camacho, 2nd degree of hypertrophy according to Camacho, 3rd degree of hypertrophy according to Camacho, 4th degree of hypertrophy according to Camacho will undergo 24-hour monitoring of oropharyngeal pH by Restech, RYAN scores upright and supine, and pH values <5.5 will be evaluated.

SUMMARY:
The study examines the severity of extraesophageal reflux using oropharyngeal pH monitoring in patients with varying degrees of lower turbinates hypertrophy.

DETAILED DESCRIPTION:
Hypertrophy of the lower turbinates causes obstruction of the nasal breathing with several health risks and a significant reduction in quality of life. Mouth breathing is non-physiological. When breathing through the mouth, the air is not purified, warmed, or humidified. This results in more frequent respiratory infections, drying of the airways, burning in the throat and causes snoring and sleep apnoea overnight. Also, nasal obstruction leads to a significant reduction in quality of life. Conservative treatment with topically applied corticosteroids is often without effect and surgical reduction of the lower turbinates under local or general anesthesia is necessary. The operation is another discomfort for the patient and is not without risks.

The pathogenesis of lower turbinates hypertrophy is multifactorial. Currently, extraesophageal reflux (EER) is considered to be a possible factor as well. The role of EER in chronic rhinosinusitis, especially in difficult-to-treat conditions, has been investigated in the past, and EER would likely be a possible co-factor. The relationship between hypertrophic lower turbinates and EER has not been studied yet.

The primary outcome/goal of the study:

To examine the severity of extraesophageal reflux using oropharyngeal pH monitoring in patients with varying degrees of lower turbinates hypertrophy.

Other goals:

* To compare extraesophageal reflux severity in patients with posterior inferior turbinate hypertrophy.
* To evaluate the difference between anterior and posterior hypertrophy of the inferior turbinates in patients with proven extraesophageal reflux.
* To evaluate the lateral difference of lower turbinates hypertrophy in patients with proven EER and in patients without proven EER.

Study protocol:

* anamnestic questionnaire (age, sex, weight, height, smoking, alcohol, reflux disease, treatment with topical corticosteroids, treatment of reflux disease)
* Reflux Symptom Index (RSI) questionnaire
* Sino-Nasal Outcome Test (SNOT 22) questionnaire
* rhinomanometry (optional - if available)
* acoustic rhinometry (optional - if available)
* olfactory questionnaire (optional - if available)
* endoscopy of the nasal cavity with evaluation:
* of the degree of hypertrophy of the lower turbinates according to Camacho, 2014 (for both turbinates separately and separately anterior and posterior half of the turbinates) (attachment 1)
* of bulky posterior inferior turbinate hypertrophy
* of reddening of the posterior ends of the lower turbinates
* of reddening of nasopharynx
* 24-hour monitoring of oropharyngeal pH by Restech, RYAN score upright and supine and pH values <5.5 will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* patients indicated for oropharyngeal pH-metry (Restech) with suspected extraesophageal reflux
* patients with 2nd - 4th degree hypertrophy of the lower turbinates (according to Camacho Classification)

Exclusion Criteria:

* patients with chronic rhinosinusitis with polyps
* patients who have had an acute upper respiratory tract infection in the last 8 weeks
* patients after previous surgery in the nasal cavity and nasopharynx
* patients after radiotherapy in the head and neck area
* non tolerance of pH catheter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Severity of extraesophageal reflux using oropharyngeal pH monitoring | 24 hours
  The primary outcome measure of the study is to examine the severity of extraesophageal reflux using oropharyngeal pH monitoring in patients with varying degrees of lower turbinates hypertrophy, assessed on the RYAN score.

CONTACTS AND LOCATIONS:
Overall Officials: Karol Zeleník, Ass.Prof.,MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (3):
- Czechia (2):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Fortmedica Prague, Prague
- Comenius University, University Hospital Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be made available to other researchers upon request.

REFERENCES:
- [Background] Camacho M, Zaghi S, Certal V, Abdullatif J, Means C, Acevedo J, Liu S, Brietzke SE, Kushida CA, Capasso R. Inferior turbinate classification system, grades 1 to 4: development and validation study. Laryngoscope. 2015 Feb;125(2):296-302. doi: 10.1002/lary.24923. Epub 2014 Sep 12. PMID 25215619
- [Background] Farmer SE, Eccles R. Chronic inferior turbinate enlargement and the implications for surgical intervention. Rhinology. 2006 Dec;44(4):234-8. PMID 17216738
- [Background] Camacho M, Zaghi S, Certal V, Abdullatif J, Modi R, Sridhara S, Tolisano AM, Chang ET, Cable BB, Capasso R. Predictors of Nasal Obstruction: Quantification and Assessment Using Multiple Grading Scales. Plast Surg Int. 2016;2016:6945297. doi: 10.1155/2016/6945297. Epub 2016 May 16. PMID 27293885
- [Background] Ayazi S, Lipham JC, Hagen JA, Tang AL, Zehetner J, Leers JM, Oezcelik A, Abate E, Banki F, DeMeester SR, DeMeester TR. A new technique for measurement of pharyngeal pH: normal values and discriminating pH threshold. J Gastrointest Surg. 2009 Aug;13(8):1422-9. doi: 10.1007/s11605-009-0915-6. Epub 2009 May 7. PMID 19421822
- [Background] Chheda NN, Seybt MW, Schade RR, Postma GN. Normal values for pharyngeal pH monitoring. Ann Otol Rhinol Laryngol. 2009 Mar;118(3):166-71. doi: 10.1177/000348940911800302. PMID 19374146
- [Background] Wiener GJ, Tsukashima R, Kelly C, Wolf E, Schmeltzer M, Bankert C, Fisk L, Vaezi M. Oropharyngeal pH monitoring for the detection of liquid and aerosolized supraesophageal gastric reflux. J Voice. 2009 Jul;23(4):498-504. doi: 10.1016/j.jvoice.2007.12.005. Epub 2008 May 12. PMID 18468849
- [Background] Zelenik K, Matousek P, Formanek M, Urban O, Kominek P. Patients with chronic rhinosinusitis and simultaneous bronchial asthma suffer from significant extraesophageal reflux. Int Forum Allergy Rhinol. 2015 Oct;5(10):944-9. doi: 10.1002/alr.21560. Epub 2015 Jun 5. PMID 26046448